CLINICAL TRIAL: NCT05210530
Title: An Open-Label, First-In-Human Study Evaluating the Safety and Tolerability of VCTX210A Combination Product in Subjects With Type 1 Diabetes Mellitus (T1D)
Brief Title: An Open-Label, FIH Study Evaluating the Safety and Tolerability of VCTX210A Combination Product in Subjects With T1D
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CRISPR Therapeutics AG (Industry)
Collaborators: ViaCyte (Industry)
Responsible Party: Sponsor
Organization: CRISPR Therapeutics (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCTX210A-101
Record Dates: First submitted 2021-12-07; First posted 2022-01-27 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Metabolic Disease; Endocrine System Diseases; Autoimmune Diseases; Immune System Diseases
Keywords: Type 1 Diabetes; T1D; Allogeneic; Combination Device; CRISPR-Cas9; Cell Therapy; T1DM; Diabetes; VCTX
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Autoimmune Diseases; Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- VCTX210A combination product (Experimental): Up to seven (7) units will be implanted
  Interventions: Combination Product: VCTX210A unit

INTERVENTIONS:
Combination Product: VCTX210A unit — CRISPR-Cas9 genetically modified PEC210A cells loaded into a delivery device

SUMMARY:
This is an open-label, multicenter, Phase 1 study evaluating the safety and tolerability of VCTX210A combination product in patients with T1D

DETAILED DESCRIPTION:
VCTX210A combination product (unit) comprises 2 components: (1) allogeneic pancreatic endoderm cells (PEC210A) genetically modified using Clustered Regularly Interspaced Short Palindromic Repeats/CRISPR-associated protein 9 (CRISPR/Cas9) to promote immune evasiveness and survival, and (2) a durable, removable, perforated device designed to deliver and retain the PEC210A cells.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of T1D for a minimum of 5 years
* Stable, optimized diabetic regimen for at least 3 months prior to enrollment

Exclusion Criteria

* Medical history of islet cell, kidney, and/or pancreas transplant
* Occurrence of 2 or more severe, unexplained hypoglycemic events within 6 months prior to enrollment
* Known causes of diabetes other than T1D
* Immunosuppressant therapy in the previous 30 days and/or requirements for chronic immunosuppressive therapy during the study
* Prior treatment with gene therapy or edited product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events with causality related to VCTX210A units and/or the surgical procedures required to implant and explant the VCTX210A units. | From implantation up to 6 months post implantation

SECONDARY OUTCOMES:
Qualitative evaluation of immune response to VCTX210A units assessed by histological staining for markers of host innate immune cells within the graft. | From implantation up to 6 months post implantation
Qualitative evaluation of immune response to VCTX210A units assessed by histological staining for markers of host adaptive immune cells within the graft. | From implantation up to 6 months post implantation
Incidence of new alloreactive antibodies found in the blood of patients post implantation. | From implantation up to 6 months post implantation
Incidence of new autoreactive antibodies found in the blood of patients post implantation. | From implantation up to 6 months post implantation
The percentage of viable graft cells per unit using immunohistochemical staining. | From implantation up to 6 months post implantation
The percentage of graft cells per unit that have differentiated into endocrine/beta cells as determined by immunohistochemical staining. | From implantation up to 6 months post implantation

CONTACTS AND LOCATIONS:
Overall Officials: Manasi Jaiman, MD, MPH, Study Director — ViaCyte; Sandeep Soni, MD, Study Director — CRISPR Therapeutics
Locations (3):
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - LMC Manna, Toronto, Ontario

REFERENCES:
- [Derived] Ellis CE, Mojibian M, Ida S, Fung VCW, Skovso S, McIver E, O'Dwyer S, Webber TD, Braam MJS, Saber N, Sasaki S, Lynn FC, Kieffer TJ, Levings MK. Human A2-CAR T Cells Reject HLA-A2 + Human Islets Transplanted Into Mice Without Inducing Graft-versus-host Disease. Transplantation. 2023 Sep 1;107(9):e222-e233. doi: 10.1097/TP.0000000000004709. Epub 2023 Aug 21. PMID 37528526